CLINICAL TRIAL: NCT00435032
Title: Early Versus Interval Appendectomy for Ruptured Appendicitis in Children. Ruptured Appendicitis Pilot Trial (RAPTOR)
Brief Title: Early Versus Interval Appendectomy for Ruptured Appendicitis in Children
Acronym: RAPTOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Martin Blakely, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R073223335
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Ruptured Appendicitis
Keywords: ruptured appendicitis; children; surgery; randomized trial
MeSH Terms: conditions — Appendicitis

ARMS (2):
- 1 (Active Comparator): Early appendectomy
  Interventions: Procedure: early appendectomy
- 2 (Active Comparator): Interval appendectomy
  Interventions: Procedure: interval appendectomy

INTERVENTIONS:
Procedure: early appendectomy — Appendectomy within 24 hours of admission
  Arms: 1
Procedure: interval appendectomy — Initial antibiotic treatment followed by appendectomy at 6-8 weeks
  Arms: 2

SUMMARY:
The purpose of this randomized trial is to compare two commonly utilized surgical treatments for children with ruptured appendicitis: early appendectomy, versus interval appendectomy. The primary outcome measure is time away from normal activities.

DETAILED DESCRIPTION:
There are two surgical treatment options for children with ruptured appendicitis. Early appendectomy is one option and typically involves removing the ruptured appendix after several hours of optimizing the patient medically with intravenous fluids and intravenous antibiotics. Another option, interval appendectomy, uses the same initial fluid and antibiotic management, but delays removing the appendix until 6-8 weeks later. The rationale for delaying the appendectomy is to perform the operation at a time when the patient is perhaps more stable and the abdominal cavity is free from contamination. Both of these treatment options are currently used by many pediatric surgeons across the United States and both appear to work well. The two treatment have never been compared in any prospective study. The primary outcome of the study is the time that a patient (and family) is away from normal activities, due to the disease and its treatment. Secondary outcome measures include complication rates, quality of life measures (SF10), hospital cost analysis, and others.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ruptured appendicitis

Exclusion Criteria:

* Inability to have usual follow up care (e.g. transient to area)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
time (days) away from normal activities (or time until returns to normal activities) | At completion of study

SECONDARY OUTCOMES:
complication rates of each treatment arm: | At completion of study
Wound infection or dehiscence | Throughout study period
Intra-abdominal abscess | Throughout study period
Requires reoperation | Throughout study period
Bowel obstruction | Throughout study period
central venous catheter-related infection | Throughout study period
interventional radiology-related complication | Throughout study period
Total hospital length of stay | At study completion
# patients with central venous line | At study completion
# with interventional radiology drainage | At study completion
# of return visits to pediatrician, ED, surgery office | At study completion
Other complication | At study completion
quality of life questionnaire (SF10) | At diagnosis, at hospital discharge, one month after diagnosis and one month after completion of all treatment
hospital costs | At study completion

CONTACTS AND LOCATIONS:
Overall Officials: Martin L Blakely, MD, Principal Investigator — University of Tennessee Health Science Center, LeBonheur Children's Medical Center; Barbara Culbreath, RN, Study Director — University of Tennessee Health Science Center, LeBonheur Children's Medical Center
Locations (1):
- LeBonheur Children's Medical Center, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Blakely ML, Williams R, Dassinger MS, Eubanks JW 3rd, Fischer P, Huang EY, Paton E, Culbreath B, Hester A, Streck C, Hixson SD, Langham MR Jr. Early vs interval appendectomy for children with perforated appendicitis. Arch Surg. 2011 Jun;146(6):660-5. doi: 10.1001/archsurg.2011.6. Epub 2011 Feb 21. PMID 21339413